CLINICAL TRIAL: NCT07085182
Title: Tislelizumab Combined With sCRT in Stage IIIB/C-IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Tislelizumab Combined With sCRT in Stage IIIB/C-IV Non-Squamous Non-Small Cell Lung Cancer：A Prospective, Single-Arm, Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zibo Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-Ethical Review -01
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: NSCLC; Tislelizumab; Chemotherapy; Hypofractionated Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): For patients with driver gene-negative stage IIIB/C-IV non-squamous non-small cell lung cancer, after 4 cycles of Tislelizumab combined with platinum-based doublet chemotherapy, if the tumor efficacy evaluation reaches SD, PR, or CR, radiotherapy will be administered to the tumor lesions combined withTislelizumab. After that, Tislelizumab maintenance therapy will be continued.
  Interventions: Drug: SBRT combined with Tislelizumab followed by Tislelizumab

INTERVENTIONS:
Drug: SBRT combined with Tislelizumab followed by Tislelizumab — SBRT:3-10Gy/F, once daily, 5 times a week; Tislelizumab(200mg,iv,q3w):Tislelizumab was added after five sessions of SBRT radiotherapy.

SUMMARY:
In clinical practice, some patients cannot tolerate concurrent chemoradiotherapy. The purpose of this study is to observe the efficacy and safety of Tislelizumab combined with platinum-based doublet chemotherapy followed by hypofractionated radiotherapy and Tislelizumab in patients with stage IIIB/C-IV non-squamous non-small cell lung cancer. This study aims to provide more treatment options for patients with locally advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
3. Patients with stage IIIB/C-IV non-squamous non-small cell lung cancer confirmed by cytology or histology;
4. Patients who have not received prior systemic therapy;

Exclusion Criteria:

1. Patients with uncontrolled autoimmune diseases;
2. Patients who have had autoimmune reactions in the past 6 months and have not improved or are unstable despite appropriate treatment, such as untreated or unstable pneumonia, thyroiditis, myocarditis, etc.;
3. Patients known to carry driver gene mutations such as EGFR mutation, ALK translocation, BRAF, ROS1, RET, MET, etc.;
4. Patients who have received prior systemic therapy, or those who have received adjuvant or neoadjuvant therapy with a recurrence time of less than 3 months from the last treatment;
5. Patients with known allergies or contraindications to the study drug or its excipients;
6. Pregnant or lactating female patients, or female patients of childbearing potential with a positive baseline pregnancy test;
7. Female patients of childbearing potential or male patients with reproductive plans who are unwilling to use effective contraception during the entire trial period and for 6 months after the end of the trial;
8. Patients whose comorbidities or other conditions may affect compliance with the protocol or are deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 30 months
  PFS is defined as the time from the first dose until the first documentation of progression or death from any cause, whichever occurs first, as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 30 months
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR), as assessed by the investigator using RECIST v1.1.
Overall Survival (OS) | Up to ~60 months
  OS is defined as the time from first dose until the date of death due to any cause
Disease Control Rate (DCR) | Up to ~24 months
  DCR is defined as the percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD), as assessed by the investigator using RECIST v1.1.
Adverse events | Through study completion, an average of 2 year
  The incidence and severity of AEs will be determined according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Zibo Municipal Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided